CLINICAL TRIAL: NCT04490850
Title: COVID-19 Seroprevalence Study in French Guiana
Acronym: EPI-COVID-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de la Guyane (Unknown); Laboratoire de biologie médicale, Institut Pasteur de la Guyane (Unknown); Laboratoire de biologie médicale de Kourou, French Guiana (Unknown); Laboratoire de biologie médicale du Centre hospitalier de Saint-Laurent du Maroni, French Guiana (Unknown); Eurofins (Industry); Centres Délocalisés de Prévention et de Soins, Centre Hospitalier Andrée Rosemon de Cayenne, Frech Guiana (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-048
Record Dates: First submitted 2020-07-28; First posted 2020-07-29 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus Infection; Severe Acute Respiratory Syndrome; SARS-CoV Infection; Covid19
Keywords: SARS-CoV-2; COVID-19; Serology; French Guiana
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Blood sample
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample

SUMMARY:
Serological surveys measuring anti-severe acute respiratory syndrome coronavirus 2 (anti-SARS-CoV-2) antibodies in the population to assess the extent of the infection and the COVID-19 immunity of the population in French Guiana.

DETAILED DESCRIPTION:
Serological surveys measuring anti-severe acute respiratory syndrome coronavirus 2 (anti-SARS-CoV-2) antibodies in the population to assess the extent of the infection and the COVID-19 immunity of the population in French Guiana.

This study is a interventional study that present minimal risks and constraints.

The results of the study will allow estimation of COVID-19 virus infection, severity and attack rates, as well as inform public health responses and policy decisions in the French Guiana territory.

ELIGIBILITY:
Inclusion Criteria:

* Person going to a prevention and care center or medical biology analysis laboratory as part of the care, regardless age, regardless of an acute or previous infection with COVID-19;
* State of health compatible with a blood sample as defined in the protocol

Exclusion Criteria:

* Inability to consent
* Person under guardianship or curatorship
* Known pathology or a health problem contraindicated with the collect of blood sample.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3541 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Measure of the COVID-19 immunity of the population | 1 year
  The COVID-19 immunity of the population will be assessed by evaluating the anti-severe acute respiratory syndrome coronavirus 2 (anti-SARS-CoV-2) antibodies

SECONDARY OUTCOMES:
Evaluation of the level of asymptomatic and pauci-symptomatic infections | 1 year
  The proportion of asymptomatic and pauci-symptomatic infections will be measured in the population

CONTACTS AND LOCATIONS:
Overall Officials: Claude Flamand, PhD, Principal Investigator — Institut Pasteur de la Guyane, Head of Epidemiology Unit
Locations (5):
- French Guiana (5):
  - Centre Hospitalier Andrée Rosemon, Cayenne
  - Laboratoire de biologie méicale, Institut Pasteur de la Guyane, Cayenne
  - Laboratoires Eurofins Guyane, Cayenne
  - Laboratoire de biologie médicale de Kourou, Kourou
  - Laboratoire de biologie médicale du Centre hospitalier de Saint-Laurent du Maroni, Saint-Laurent-du-Maroni